CLINICAL TRIAL: NCT04773327
Title: A Multicenter, Randomized Controlled, Open Clinical Study of the Efficacy and Safety of PEG-rhG-CSF in the Prevention of Neutropenia After Chemotherapy in Patients With Gynecological Malignancies
Brief Title: Efficacy and Safety of PEG-rhG-CSF in the Prevention of Neutropenia After Chemo in Pts With Gynecological Malignancies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xiaohua Wu MD (Other)
Responsible Party: Sponsor-Investigator, Xiaohua Wu MD, director of gynecologic oncology, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MA-GynC-II-001
Record Dates: First submitted 2021-02-02; First posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Gynecologic Malignant Tumor
Keywords: neutropenia
MeSH Terms: conditions — Neutropenia | interventions — pegylated granulocyte colony-stimulating factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PEG-rhG-CSF prevention (Experimental): Mecapegfilgrastim subcutaneous injection, 6mg, 24-48h after the end of antitumor drug administration in each chemotherapy cycle,
  Interventions: Other: Mecapegfilgrastim Injection
- non-prevention (No Intervention): Only close monitoring after chemotherapy

INTERVENTIONS:
Other: Mecapegfilgrastim Injection — 24-48h after the end of antitumor drug administration in each chemotherapy cycle, Mecapegfilgrastim was injected subcutaneously, 6mg/ time, once/cycle
  Other Names: PEG- rhg - csf
  Arms: PEG-rhG-CSF prevention

SUMMARY:
This study is a multi-center, forward-looking, open, randomized, controlled clinical trial. This study aims to analyze the effects of Mecapegfilgrastim Injection prevention versus non-prevention for neutropenia in ovarian cancer, cervical cancer, endometrial cancer patients after chemical therapy.

Patients are randomized into study group and control group. All patients receive PTX+platinum chemotherapy of 3 weeks. In study group, patients accept PEG-rhG-CSF 24-48 hours from the chemotherapy. While the control group patients are only observed closely. Patient receive three courses of treatment.

The primary end is the incidence of 3/4 level neutropenia in three courses of chemotherapy.

The secondary ends include: the incidences and duration of neutropenia in every course of chemotherapy, the incidences of FN in three courses and every course of chemotherapy, the incidences of infection in three courses and every course of chemotherapy, the delay time of the next cycle of chemotherapy due to FN or infection, the RDI of the second and third cycles of chemotherapy, adverse events related to G-CSF, quality of life, cost of medicine and admitting.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-70
* Weight ≥45 kg
* ≤2 lines chemotherapy or postoperative adjuvant chemotherapy patients with cervical cancer, ovarian cancer and endometrial cancer
* Receive paclitaxel combined with platinum three weeks per cycle of chemotherapy
* With an Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1
* Expected survival time of > 3 months
* Main organ functions meet the following criteria:

  1. Hb≥75g/L; WBC≥3.0×109/L; ANC≥1.5×109/L; PLT≥80×109/L;
  2. APTT-ULN≤10s; PT-ULN≤3s; TT-ULN≤3s;
  3. ALT≤2.5×ULN; AST≤2.5×ULN; TBIL≤2.5×ULN;
  4. BUN≤1.5×ULN; Cr≤1.5×ULN; UA≤1.5×ULN；Creatinine clearance≥40mL/min;
  5. without obvious cardiac dysfunction
* Provided consent for participation

Exclusion Criteria:

* With uncontrollable infections or receive systemic antibiotics within 72 hours prior to chemotherapy
* Pregnant or lactating women
* Received bone marrow or hematopoietic stem cell transplantation within the past 3 months
* Concurrent chemoradiotherapy
* Presence of hematological disorders: systemic lupus erythematosus, sjogren's syndrome, rheumatic autoimmune disease, mixed and hoof tissue disease, autoimmune hemolytic anemia, leukopenia , chronic granulocyte leukemia, bone marrow dysplasia syndrome, aplastic anemia, congenital and idiopathic neutropenia, myelodysplastic syndrome, cyclic neutropenia, primary and secondary thrombocytopenic purpura, etc
* Presence of risk of thrombus or high risk of clotting
* Presence of psychosis, neurological disease or brain metastases from tumors
* Presence of uncontrollable complicated disease including symptomatic congestive heart failure, uncontrollable hypertension, unstable angina pectoris, active peptic ulcer, or hemorrhagic disease
* Presence of uncontrollable infectious diseases, active viral hepatitis, tuberculosis, HIV
* Allergic to recombinant human granulocyte stimulating factor or other biological products of E. coli origin
* Received clinical trials within 1 month prior to enrollment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of third/fourth level neutropenia | three months
  Incidence of third/fourth level neutropenia during three cycles chemotherapy

SECONDARY OUTCOMES:
Incidence of febrile neutropenia | three months
  Incidence of febrile neutropenia during every cycle chemotherapy
The duration time of third/fourth level neutropenia | three months
  The duration time of third/fourth level neutropenia during three cycles chemotherapy
Incidence of infection | three months
  Incidence of third/fourth level neutropenia during three cycles chemotherapy
delay time of chemotherapy | three months
  The delay time of the next cycle of chemotherapy due to FN or infection
RDI of chemotherapy | three months
  Relative dose intensity of the second and third chemotherapy
Adverse events | three months
  Incidence of adverse events related to granulocyte colony stimulating factor according to common Terminology Criteria for Adverse Events (CTCAE) v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohua Wu, MD&PHD, Principal Investigator — director of gynecologic oncology
Locations (1):
- No. 270, Dongan Road, Xuhui District, Shanghai, China, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
data is available per require after approved by ethics broad